CLINICAL TRIAL: NCT04330482
Title: Translating a Dementia Caregiver Intervention Into a Mobile Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: University of Rhode Island (Other)
Responsible Party: Principal Investigator, Geoffrey Tremont, Director of Neuropsychology, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R21AG064410-01 (NIH)
Record Dates: First submitted 2020-03-19; First posted 2020-04-01 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Dementia; Alzheimer Disease; Caregiver Burnout
Keywords: MobileHealth; Caregiving; Dementia; Alzheimer Disease
MeSH Terms: conditions — Dementia; Alzheimer Disease; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: A full-scale randomized, controlled trial: 20 participants will be randomized to receive a tablet pre-loaded with a list of internet links relevant to dementia caregiving and 20 participants will be randomized to receive a tablet pre-loaded with the CARE-Well App. Both groups will be instructed to use their tablets at least 4 times per week for 3 months.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet Links (Other): A tablet pre-loaded with a list of internet links relating to dementia caregiving that participants will be instructed to use at least 4 times weekly for 3 months.
  Interventions: Behavioral: Internet Links
- CARE-Well App (Experimental): A tablet pre-loaded with the CARE-Well app that participants will be instructed to use at least 4 times weekly for 3 months.
  Interventions: Behavioral: CARE-Well App

INTERVENTIONS:
Behavioral: CARE-Well App — Participants randomized into this group will be instructed to use the CARE-Well App at least 4 times per week.
  Arms: CARE-Well App
Behavioral: Internet Links — Participants randomized into this group will be instructed to use a computer tablet pre-loaded with a list of internet links relevant to dementia caregiving at least 4 times per week.
  Arms: Internet Links

SUMMARY:
The overall goal of this development project is to combine elements of two efficacious interventions into a mobile health (mHealth) App for informal dementia caregivers. The investigators will conduct a 3-month feasibility trial of the newly-developed CARE-Well App in 40 dementia caregivers to establish acceptability and feasibility of the intervention, study procedures, and outcome measures.

DETAILED DESCRIPTION:
Caring for a person with dementia is a highly stressful activity and is associated with negative physical and mental health consequences, including increased risk of depression and worse reported health-related quality of life. The proposed project aims to develop and translate an evidence-based, multi-component intervention into a mHealth App that has the potential to increase dementia caregivers' access to support and care.

The investigators will conduct a feasibility trial, in which 40 dementia caregivers will be randomized to receive a computer tablet preloaded with the CARE-well App or preloaded with internet links relevant to dementia and caregiving. Paper outcome measures will be assessed at baseline and end of intervention (3 months) during each study visit. To measure sustainability of the App, the first 10 caregivers from each group will be offered the tablets for an additional month to monitor usage of the App outside the formal trial. The goal of this aim is to determine feasibility of the intervention, study procedures, and outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Adequate English-speaking and reading skills
* Provide at least 4 hours of supervision per day for the care recipient (either directly or by telephone)
* Live in the community (either with the care recipient or without)
* Have provided supervision/ assistance for at least 6 months prior to study enrollment and have no plans to place care recipient in long term care or to end their role as caregiver within 6 months of study enrollment.
* Report some degree of distress associated with caregiving
* Access to Wifi at home

Exclusion Criteria:

* Major acute medical illness
* Severe mental illness (e.g. bipolar, schizophrenia)
* Diagnosed cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Tremont, PhD, Principal Investigator — Rhode Island Hospital; Kunal Mankodiya, PhD, Principal Investigator — University of Rhode Island
Locations (2):
- United States (2):
  - University of Rhode Island, Kingston, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Internet Links | CARE-Well App
Started | 20 | 20
Completed | 18 | 16
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Internet Links | CARE-Well App | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 6 | 16
  >=65 years | 10 | 14 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.70 (8.15) | 64.05 (12.43) | 66.38 (10.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 18 | 20 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 19 | 19 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Depression [Mean (Standard Deviation); unit: units on a scale] — Center for Epidemiologic Studies- Depression Scale; scores range from 0-30; higher scores reflect greater depression
  units on a scale | 12.95 (8.02) | 13.55 (9.69) | 13.25 (9.69)

OUTCOME MEASURES:

1. Primary Outcome: Randomization
Description: Percentage of participants who decline participation because of randomization.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Internet Links | CARE-Well App
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

2. Primary Outcome: Study Enrollment Rate and Retention
Description: Percentage of participants enrolled and who remain enrolled for the duration of the study.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Internet Links | CARE-Well App
Number analyzed (Participants) | 20 | 20
Participants | 18 | 16

3. Primary Outcome: Intervention Adherence
Description: Percentage of participants who used the internet links or the app for the 3-month intervention period.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Internet Links | CARE-Well App
Number analyzed (Participants) | 18 | 16
Participants | 18 | 16

4. Primary Outcome: Timing of Assessments
Description: Percentage of participants who completed assessments at baseline and follow-up within two weeks of enrollment or completion of the study.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Internet Links | CARE-Well App
Number analyzed (Participants) | 18 | 16
Participants | 18 | 16

5. Primary Outcome: Completion Rates
Description: Percentage of participants who completed the intervention.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Internet Links | CARE-Well App
Number analyzed (Participants) | 20 | 20
Participants | 18 | 16

6. Primary Outcome: Interest in Continuation of Tablet/App Use After Formal Trial
Description: Percentage of participants in a subset of caregivers (10 from each group) interested in continuing to use tablet/App use after formal trial as an estimate of sustainability.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Internet Links | CARE-Well App
Number analyzed (Participants) | 10 | 10
Participants | 10 | 10

7. Primary Outcome: App Technology Satisfaction
Description: Percentage of participants satisfied or very satisfied with App technology.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Internet Links | CARE-Well App
Number analyzed (Participants) | 18 | 16
Participants | 13 | 12

8. Primary Outcome: App Content Satisfaction
Description: Percentage of participants satisfied or very satisfied with App content.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Internet Links | CARE-Well App
Number analyzed (Participants) | 18 | 16
Participants | 13 | 11

9. Secondary Outcome: Center for Epidemiologic Studies Depression Scale
Description: Depression scale; 0-30 points; higher scores indicate worse outcome.
Time Frame: Baseline and immediately Post-Intervention at 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Internet Links | CARE-Well App
Number analyzed (Participants) | 18 | 16
units on a scale
  Baseline | 13.29 (7.88) | 13.94 (12.19)
  Post-Intervention | 16.71 (8.36) | 17.38 (11.67)

10. Secondary Outcome: Zarit Burden Interview
Description: Caregiver burden scale; 0-88 points; higher scores indicate worse outcome.
Time Frame: Baseline and immediately Post-Intervention at 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Internet Links | CARE-Well App
Number analyzed (Participants) | 18 | 16
units on a scale
  Baseline | 55.53 (9.82) | 56.56 (14.40)
  Post Intervention | 58.11 (10.93) | 57.56 (13.22)

11. Secondary Outcome: Revised Memory and Behavior Problem Checklist
Description: Caregiver reaction to problem behaviors; range 0-96 Higher scores indicate worse outcomes.
Time Frame: Baseline and immediately Post-Intervention at 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Internet Links | CARE-Well App
Number analyzed (Participants) | 18 | 16
units on a scale
  Baseline | 22.88 (7.90) | 22.00 (8.61)
  Post Intervention | 18.10 (10.56) | 11.56 (16.91)

12. Secondary Outcome: Desire to Institutionalize Scale
Description: Caregiver desire to institutionalize care recipient; 0-7 points; high scores indicate worse outcome (or stronger desire to institutionalize).
Time Frame: Baseline and immediately Post-Intervention at 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Internet Links | CARE-Well App
Number analyzed (Participants) | 18 | 16
units on a scale
  Baseline | 0.82 (1.24) | 1.38 (1.45)
  Post Intervention | 1.12 (1.54) | 1.94 (2.29)

ADVERSE EVENTS:
Time Frame: 3 months for each participant
Arm/Group | Internet Links | CARE-Well App
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/82/NCT04330482/Prot_000.pdf